CLINICAL TRIAL: NCT02607319
Title: Effect of Low Molecular Weight Heparin (Bemiparin) on Implantation Rate in Patients With Recurrent Implantation Failure Undergoing IVF/ICSI - A Prospective Randomized Clinical Trial
Brief Title: Low Molecular Weight Heparin to Improve Pregnancy Outcome in Patients With Recurrent Implantation Failure
Acronym: BRIF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Johnny Awwad, Professor of Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AmericanUBMCRIF
Record Dates: First submitted 2015-11-11; First posted 2015-11-18 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Sterility
Keywords: Recurrent Implantation Failure; Implantation; low molecular weight heparin; In vitro Fertilization; Assisted Reproductive Technology; Pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Low molecular weight heparin (Experimental): Bemiparin sodium 3,500 IU anti Xa/0.2 ml solution (Hibor; Laboratories Rovi Pharmaceuticals) for injection in pre-filled syringes.
  Interventions: Drug: Bemiparin sodium
- No intervention group (No Intervention): Control group receiving standard care.

INTERVENTIONS:
Drug: Bemiparin sodium — Bemiparin sodium 3,500 IU will be started on the evening of the same day of embryo transfer and until the day of pregnancy test. If the test is positive, Bemiparin will be discontinued by the end of the 12th week of gestation.
  Other Names: Hibor
  Arms: Low molecular weight heparin

SUMMARY:
The objective of this study is to determine the effect of Bemiparin, a low molecular weight heparin, on implantation rate in women with unexplained recurrent implantation failure undergoing IVF/ICSI treatment.

DETAILED DESCRIPTION:
Recurrent implantation failure (RIF), defined as failure of conception following three or more consecutive In Vitro Fertilization (IVF) cycles despite the transfer of good quality embryos, is a major cause of distress amongst infertile couples. While factors underlying implantation failure are many, most cases remain unexplained. In order to improve pregnancy outcomes and delivery rates in women with unexplained RIF, various investigational treatments have been proposed.

The investigators propose a prospective controlled randomized comparative study to evaluate the effect of Bemiparin on implantation rates in women with unexplained RIF. A total of 200 patients will be recruited and randomized between two groups. The study group will receive Bemiparin plus standard care; while the control group will receive only standard care. Treatment will start on the day following embryo transfer and will be continued until 12 weeks gestation in the event of pregnancy.

The primary objective is to determine the effect of Bemiparin on implantation rate in women with unexplained recurrent implantation failure.

ELIGIBILITY:
Inclusion Criteria:

* History of three or more consecutively failed In Vitro Fertilization (IVF) cycles after embryo transfer.
* Normal uterine cavity (as assessed by hysteroscopy or HSG).
* Normal hormonal investigation: TSH, PRL, FBS.
* Normal acquired/inherited thrombophilia profile: LAC, ACA IgG/IgM, Prot S, Antithrombin III, beta-2 glycoprotein, Factors V, II, MTHFR.
* Normal semen analysis and mild/moderate male factor (Total motile sperm count > 5 million/ml and/or normal WHO morphology >20%.
* Patient provides written informed consent.

Exclusion Criteria:

* Evidence of low ovarian reserve by at least one of the following: AMH ≤ 1,5 ng/mL and/or basal CD 3 FSH ≥ 10 mIU/mL and/or basal CD 3 Estradiol ≥ 60 ng/mL and/or previous egg collection yield ≤ 3 oocytes.
* Preexisting medical condition (thyroid disease, diabetes mellitus, hypertension, pulmonary conditions, cardiac condition…).
* Severe male factor infertility (Total motile sperm count < 5 million/ml and/or normal WHO morphology <20%).
* Hypersensitivity to Heparin or its derivatives.
* Acquired thrombophilia.
* Active hemorrhage or increased risk of bleeding due to impairment of homeostasis.
* Severe impairment of liver or pancreatic function.
* Severe renal insufficiency (Creatinine Clearance < 30 ml/min).
* Injuries to or operations on the central nervous system, eyes and ears within the last 2 months.
* Disseminated Intravascular Coagulation (DIC) attributable to heparin-induced thrombocytopenia.
* Acute bacterial endocarditis and endocarditis lenta.
* Any organic lesion with high risk of bleeding (e.g.: active peptic ulcer, hemorrhagic stroke, cerebral aneurysm or cerebral neoplasms).

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Implantation rate (%) | Vaginal ultrasound at 8 weeks gestation
  Number of intrauterine gestational sacs observed by transvaginal ultrasonography divided by the number of transferred embryos

SECONDARY OUTCOMES:
Live birth rate (%) | Time of delivery up to 42 weeks gestation
  birth of live born
Ongoing pregnancy rate (%) | Vaginal ultrasound at 20 weeks of gestation
  Fetal heart beat seen by ultrasound at 20 weeks gestation
Clinical pregnancy rate (%) | Vaginal ultrasound at 8 weeks gestation
  Fetal heart beat seen by ultrasound at 8 weeks gestation
Total pregnancy rate (%) | Up to 15 days from oocyte collection
  Positive hCG titer

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Awwad, MD, Principal Investigator — AUBMC
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided